CLINICAL TRIAL: NCT00002144
Title: The Pilot Study of Foscarnet Cream in the Treatment of Mucocutaneous Herpes Simplex Virus Infections in Immunocompromised Patients Unresponsive to Acyclovir Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astra USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 240A; 92-FT-57
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: Herpes Simplex; Foscarnet; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
PRIMARY: To evaluate the clinical activity of foscarnet cream on the index lesion of mucocutaneous herpes simplex virus (HSV) infections in immunocompromised patients previously unresponsive to acyclovir treatment.

SECONDARY: To evaluate the clinical activity and virologic activity of foscarnet cream on all treated lesions in this patient population. To evaluate the local tolerance and side effects of treatment with foscarnet cream in this patient population.

DETAILED DESCRIPTION:
Patients receive topical applications of one percent foscarnet cream five times daily for up to 6 weeks; those who show no evidence of epithelialization of the index lesion after 3 or more weeks are removed from study and offered intravenous foscarnet. Patients who show a good response to topical foscarnet cream at the end of 6 weeks may continue receiving treatment at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Ganciclovir (provided drug was administered for at least 14 days prior to study entry, and the HSV isolate exhibits resistance against acyclovir).
* Other medication considered necessary for patient's welfare, at the discretion of the investigator.

Patients must have:

* HIV infection or AIDS.
* Mucocutaneous HSV infection with at least one clinically evaluable lesion.
* Prior acyclovir without clinical benefit.
* Life expectancy of at least 3 months.
* Consent of parent or guardian if less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity to the study drug.
* Any medical, psychiatric, or other condition that would preclude study compliance.
* Incapable of self administration of medication or presence of a care provider administering medication.

Concurrent Medication:

Excluded:

* Intravenous foscarnet for current episode of HSV.
* Acyclovir, interferon, or any investigational drug that might have anti-HSV activity (e.g., 256U87, HPMPC, BVDaraU, trifluridine).

Patients with the following prior condition are excluded:

Previous participation in the study.

Prior Medication:

Excluded:

* Intravenous foscarnet within 2 months prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12

CONTACTS AND LOCATIONS:
Overall Officials: Hardy WD, Study Chair
Locations (8):
- United States (8):
  - CARE Ctr / UCLA Med Ctr, Los Angeles, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - South Miami Hosp, Miami, Florida
  - Dr Thomas Klein, Chicago, Illinois
  - Bellevue Hosp Ctr, New York, New York
  - Univ Hosps of Cleveland, Cleveland, Ohio
  - Roger Williams Med Ctr, Providence, Rhode Island
  - Milwaukee County Med Complex, Milwaukee, Wisconsin

REFERENCES:
- [Background] Hardy D, Javaly K, Wohlfeiler M, Kalayjian R, Klein T, Bryson Y, Graford K, Martin-Munley S. Phase I, pilot study of the safety and efficacy of foscarnet (PFA) cream for treatment (Rx) of acyclovir-unresponsive (ACV-R) herpes simplex (HSV). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:83